CLINICAL TRIAL: NCT03308604
Title: Phase I Study of AGuIX Gadolinium-based Nanoparticles in Combination With Chemoradiation and Brachytherapy in Locally Advanced Cervical Cancer
Brief Title: AGuIX Gadolinium-based Nanoparticles in Combination With Chemoradiation and Brachytherapy
Acronym: NANOCOL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-005127-83; 2016/2508 (Other: CSET number)
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Gynecologic Cancer
MeSH Terms: interventions — AGuIX; Drug Therapy; Cisplatin

STUDY DESIGN:
Intervention Model Description: This is a phase 1 clinical trial evaluating the safety, tolerability of escalating doses of AGuIX-NP in combination with radiation and cisplatin in patients with locally advanced cervical cancer. Dose escalation will be conducted using the modified toxicity probability interval (mTPI) method. Three dose levels of intravenous AGuIX nanoparticles will be explored: 20mg/kg (level -1), 30 mg/kg (level 1) and 50 mg/kg (level 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with locally advanced cervical cancer (Experimental)
  Interventions: Drug: Polysiloxane Gd-Chelates based nanoparticles (AGuIX); Radiation: External beam radiotherapy (EBRT); Radiation: Uterovaginal brachytherapy; Drug: Chemotherapy (cisplatin)

INTERVENTIONS:
Drug: Polysiloxane Gd-Chelates based nanoparticles (AGuIX) — Three intravenous injections of AGuIX will be delivered.
  The first injection of AGuIX will be delivered intravenously the 1st day and the 11th day of EBRT. The first injection will be preceded with an MRI (unenhanced T1 and T2 sequences) then followed with another MRI performed 4 hours later, to monitor tumor uptake.
  Irradiation will be performed after the second MRI.
  The second injection will be followed by an MRI 4 hours later.
  The third injection will be delivered intravenously the day of the brachytherapy procedure. Intravenous hydration will be performed during all brachytherapy courses to ensure AGuIX clearance.
  Up to three dose levels may be explored: 20mg/kg (level -1), 30 mg/kg (level 1) and 50 mg/kg (level 2). The starting dose level will be 30mg/kg.
Radiation: External beam radiotherapy (EBRT) — to the pelvis, with intensity modulated technique: 45 Gy in 5 weeks, with integrated boost to 55 - 57.5 Gy in case of macroscopic lymph node metastases
Radiation: Uterovaginal brachytherapy — 15 Gy (maximal interval between EBRT and brachytherapy: 14 days).
Drug: Chemotherapy (cisplatin) — Concomitant weekly intravenous cisplatin 40 mg/m2 will be delivered (total 5 cycles).

SUMMARY:
This is a phase 1 clinical trial evaluating the safety, tolerability of escalating doses of AGuIX-NP in combination with radiation and cisplatin in patients with locally advanced cervical cancer. Dose escalation will be conducted using the modified toxicity probability interval (mTPI) method.

Three dose levels of intravenous AGuIX nanoparticles will be explored: 20mg/kg (level -1), 30 mg/kg (level 1) and 50 mg/kg (level 2).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed cancer of the uterine cervix: squamous cell carcinoma or adenocarcinoma stage IB2-IVA according to the International Federation of Gynecology and Obstetrics classification, regardless of the pelvic lymph node stage. No evidence of metastatic disease. Primary staging should include: clinical examination, Pelvic MRI and 18-FDG PET. A coelioscopic para-aortic lymph node staging should be done in patients without para-aortic lymph node uptake to guide radiotherapy fields in the situation of pelvic lymph node metastases. If there is no pelvic lymph node metastases, para-aortic lymph node dissection is optional.
2. ECOG performance status 0-1.
3. Age between 18 - 70 years.
4. Neutrophils > 2000/mm^3.
5. Hemoglobin > 9 g/L after transfusion if necessary.
6. Platelets > 100,000/mm^3.
7. Creatinine < 1.5 upper limit of normal or calculated creatinine clearance (Cockcroft-Gault Formula) ≥ 60 mL/min.
8. Liver function (GOT, GPT, alkaline phosphatase and bilirubin) < 1.5 upper limit of normal.
9. Cardiovascular: no clinically relevant cardiovascular disease, no congestive heart failure, no symptomatic coronary artery disease, no poorly controlled cardiac arrhythmia, no myocardial infarction within the past year.
10. Gastrointestinal: no active inflammatory bowel disease, no lack of physical integrity of the upper gastrointestinal tract, no malabsorption syndrome.
11. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to initiation of treatment.
12. Proteinuria < 2 g/L (200mg/dL) and creatinine clearance ≥ 60 mL/min.
13. Signed informed consent after informing the patient.
14. Patient affiliated to a social security regimen or beneficiary of the same.

Exclusion Criteria:

1. Other histological types of cervical cancer than those listed in the inclusion criteria or stage IVB.
2. History of cancer other than basal cell carcinoma within five past years.
3. Prior treatment with radiotherapy, chemotherapy, targeted therapy or immune therapy for cervical cancer or for any cancer within five past years.
4. Prior pelvic radiotherapy or prior surgical treatment for cervical cancer (excluding diagnostic conisation).
5. Pregnancy or breastfeeding.
6. Obesity (Body Mass Index > 30).
7. History of prior or current psychiatric illness.
8. Nephropathy, regardless of the grade.
9. Peripheral neuropathy ≥ grade 2.
10. Patients with pre-existing hearing impairments.
11. Active infection or other serious underlying pathology that could prevent the patient from receiving the treatment (especially liver or heart conditions).
12. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
13. Positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
14. Inclusion in another clinical trial protocol with an experimental molecule (during this study or within 5 years prior to enrollment).
15. Unable to undergo the follow-up required by study for geographical, social or psychological reasons.
16. Contra-indication for Magnetic Resonance Imaging enhanced with gadolinium and/or any contra-indication to the use of cisplatin.
17. History of allergic reaction to cisplatin or other platinum containing compounds.
18. Concurrent administration of yellow fever vaccine.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynecologic Cancer
Enrollment: 18 (Estimated)
Dates: Start 2018-05-17 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Day 84 after inclusion
Recommended Phase 2 Dose (RP2D) | Day 84 after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Cyrus CHARGARI, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (2):
- France (2):
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhône
  - Gustave Roussy, Villejuif, Val De Marne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maury P, Mondini M, Chargari C, Darricau A, Shahin M, Ammari S, Bockel S, Genestie C, Wu TD, Lux F, Tillement O, Lacombe S, Deutsch E, Robert C, Porcel E. Clinical transfer of AGuIX(R)-based radiation treatments for locally advanced cervical cancer: MR quantification and in vitro insights in the NANOCOL clinical trial framework. Nanomedicine. 2023 Jun;50:102676. doi: 10.1016/j.nano.2023.102676. Epub 2023 Apr 20. PMID 37084803